CLINICAL TRIAL: NCT05090774
Title: Integrating Fall Prevention Balance Exercises Into a Program for Older Adults With Peripheral Artery Disease (PAD): A Mixed Methods Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SON-2021-30171
Record Dates: First submitted 2021-10-06; First posted 2021-10-25 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Fall; Fall Injury; Peripheral Artery Disease; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Exercise Therapy (SET) Plus Balance Exercises (Experimental): Intervention meetings surrounding supervised exercise therapy (SET) with the addition of the adapted Otago Exercise Program (OEP) will occur individually with participants in a 1:1 format once per week for 30 minutes over 8 weeks. Additionally, participants will be encouraged to practice exercises at home at least 2 additional days between intervention meetings using visual handouts (up to 7 times/week total, approximately 140 minutes/week).
  Interventions: Behavioral: Adapted Otago Exercise Program (OEP)
- Supervised Exercise Therapy (SET) Only (No Intervention): Intervention meetings surrounding supervised exercise therapy (SET) will occur individually with participants in a 1:1 format once per week for 30 minutes over 8 weeks. Additionally, participants will be encouraged to practice exercises at home at least 2 additional days between intervention meetings using visual handouts (up to 7 times/week total, approximately 140 minutes/week).

INTERVENTIONS:
Behavioral: Adapted Otago Exercise Program (OEP) — A modified version of the 8- week evidence-based Otago Exercise Program (OEP), adapted for integration into supervised exercise therapy (SET). The OEP exercises will include 12 static and dynamic standing balance movements (knee bends, backwards walking, walking and turning, sideways walking, tandem stance, tandem walk, one leg stand, heel walking, toe walking, heel-toe walking backwards, sit to stand, stair walking). The OEP also contains additional behavior change techniques embedded within the intervention protocol (i.e. feedback on behavior, self-monitoring of behavior, biofeedback).
  Arms: Supervised Exercise Therapy (SET) Plus Balance Exercises

SUMMARY:
The overarching objective of this study is to improve fall prevention efforts in community-dwelling older adults with peripheral artery disease (PAD) to reduce falls. To accomplish this, the investigators will conduct a feasibility study and pilot the addition of a balance exercise component to existing supervised exercise therapy (SET) programs for PAD. This intervention may be an effective way to help older adults with PAD self-manage their leg pain and walking impairments as well as fall risk. The long-term goal of this research is to reduce morbidity and mortality associated with falls in older adults with symptomatic PAD through the development and evaluation of a balance intervention component implemented within existing exercise programs. Findings from this research may also be translated to the implementation of disease management programs for other chronic conditions associated with fall risk. The rationale for this research is to determine improve disease-specific, comprehensive and fall prevention strategies for older adults with PAD.

DETAILED DESCRIPTION:
Falls are a growing public health concern as the proportion of aging adults will continue to increase in the coming years and the prevalence of falls is high. Older adults with PAD have previously demonstrated impaired static balance, higher prevalence of history of stumbling/unsteadiness (41%) and falling (26%), and abnormal balance using computerized dynamic posturography compared to non-PAD controls. Adults with symptomatic PAD also demonstrate LE weakness and gait deficiencies due to impaired muscle power and biomechanics. While still unspecified, muscle weakness and ischemic neuropathy could partially explain the etiology for impaired balance in those with PAD. Other potential associations with increased fall risk in PAD may include claudication, limited physical activity, and poor LE function. Through expansion of disease-specific knowledge related to fall prevention interventions in older adults with PAD, healthcare providers may find that targeted balance screening and interventions to improve balance and strength are essential to disease management and the prevention of disability. The proposed study is innovative as it is the first balance intervention study in PAD and uses an explanatory sequential mixed methods design. Given the known associations between PAD and balance, in addition to morbidity and mortality associated with falls in the general population of older adults, the contribution of this knowledge is unique in that it will improve understanding of interventional study designs, leading to future revisions in prevention strategies for this sub-group.

Findings from a recent systematic review of fall prevention interventions for community-dwelling older adults with chronic conditions suggest that the stage of intervention development primarily lies within efficacy-based RCTs that focus on internal validity, which limits the generalizability of these intervention effects for varying contexts. Most of these interventional studies did not report detail related to adoption and maintenance, such as recruitment of participants from the target populations and intervention adoption by staff, which are critical to understanding how to implement these interventions in clinical settings. There was also a lack of qualitative research methods use across the studies, which limits the understanding of participants' acceptability and perceived intervention effects. Most of these trials were conducted in controlled research setting environments adjacent to, but not integrated within, clinical practice settings without staff involvement, which impacts the adoption of these programs. While all of the studies in the review included targeted, individuals, and moderately challenging balance exercises (some with additional strength and aerobic training components), the dosing of balance exercises was not sufficient to meet the exercise duration recommendations over the intervention period. Due to the stage of development, it is challenging to evaluate the long-term implementation and public impact of these interventions with delivery performed by clinicians and community partners who have direct contact with this target population. Despite the inextricable relationships between fall risk and PAD, self- management interventions for fall risk and PAD are currently not integrated into PAD treatment. Often, interventions for self-management of chronic conditions and fall prevention are delivered separately. Given the complexity, time, and effort required for PAD self-management programs, a separate stand- alone program for fall prevention exercises is unlikely due to its added burden on patients. Thus, there is a need to explore the feasibility of integrating evidence- based fall prevention exercises into existing PAD programs. Some researchers have investigated the integration of rehabilitation programs and fall prevention in patients with chronic obstructive pulmonary disease, where balance exercises were delivered as part of either outpatient and inpatient pulmonary rehab. Although balance training has not been implemented as a standard treatment for PAD subgroups, there is potential for its addition to established PAD programs. Many older adults with PAD participate in outpatient supervised exercise therapy (SET) walking programs, which are the most effective non-invasive method to mitigate claudication and improve walking function in adults with PAD. In addition to mitigating fall risk, the combined balance training within SET programs also has potential to improve patient outcomes. Balance training could be an adjunct to the SET standard of care, which is designed to improve claudication symptoms and address walking function. Although intermittent treadmill walking is the optimal mode to maximize benefits from exercise training for PAD, it is often contraindicated or refused due to poor balance. As walking demands adequate balance, LE strength, and endurance, individuals with poor postural control may benefit from improving their balance prior to or during the initiation of walking exercise to manage their vascular disease. Thus, the simultaneous learning and mastering of balance exercises to reduce fall risk may enable successful participation in treadmill walking, thus maximizing the benefits gained from SET.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in supervised exercise therapy (SET)
* One or more fall risk factors as determined by CDC STEADI fall risk screener

  * One or more falls in the last year
  * Unsteadiness when standing or walking
  * Worries about falling
* Have symptomatic peripheral artery disease (PAD) with objective diagnosis (ABI less than or equal to 0.90 or previous revascularization)

Exclusion Criteria:

* Formal diagnosis of neurocognitive impairment or <3 on Callahan 6-Item Screener
* Current uncontrolled vestibular dysfunction (e.g. Meniere's Disease, benign paroxysmal positional vertigo)
* Participants who self-report the following symptoms will require clearance from a primary provider (as guided by the Exercise and

Screening for You Questionnaire):

* Pain, tightness or pressure in chest during physical activity (walking, climbing stairs, household chores, similar activities) that have not been checked and/ or treated by a healthcare provider
* Current dizziness that have not been checked and/ or treated by a healthcare provider
* Current, frequent falls that have not been checked and/ or treated by a healthcare provider

  * Other clinically significant disease that is, in the opinion of the study team, not stabilized or may otherwise confound the results of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Mini-Balance Evaluation Systems Test Score | Baseline and 8 weeks
  The Mini-Balance Evaluation Systems Test consists of 14 items with total scores ranging from 0-28. Higher scores indicate better balance performance. Balance will be evaluated pre- and post-intervention.

SECONDARY OUTCOMES:
Percent Target Recruitment | Baseline and 8 weeks
  The percent of target recruitment achieved will be assessed pre- and post-intervention as a measure of demand.
Rate of Participants Enrolled Per Month | 8 weeks
  Enrollment rates per month will be reported as participants per month as a measure of demand.
Percent of Participants that Complete 8-Week Intervention | 8 weeks
  The percent of participants that complete the 8-week intervention out of total participants will be reported as a measure of retention and acceptance.
Satisfaction Questionnaire Score | 8 weeks
  Satisfaction with and evaluation of the program will be assessed via a 5-item Likert scale ranging from 'Strongly Disagree' to 'Strongly Agree', where higher scores indicate greater satisfaction.
Interventions Attended | 8 weeks
  Attendance will be measured as the average number of intervention sessions attended across participants and reported as a number of sessions.
Adherence to Home-Based Balance Exercises | 8 weeks
  Intervention fidelity will be measured via adherence to home-based balance exercises and reported as the average number of days that participants exercised at home per week. Adherence will be assessed weekly via an exercise tracker.
Change in Timed Up and Go (TUG) Test Score | Baseline and 8 weeks
  The TUG test measures the time it takes to stand from a chair, walk 10 feet, turn around, walk to the chair, and sit and will be reported in seconds. TUG test will be assessed pre- and post-intervention.
Change in Short Performance Physical Battery (SPPB) Score | Baseline and 8 weeks
  The SPPB is reported as a score on 5 balance, strength, and walking tests that evaluate lower extremity function. The range of summed scores is 0-12, where 12 indicates better lower extremity function. The SPPB will be assessed pre- and post-intervention.
Fall Rates Per Month | 8 weeks
  The average monthly rate of self-reported falls over the intervention period will be reported as falls per month.
Change in Falls Efficacy Scale-International Score | Baseline and 8 weeks
  The Falls Efficacy scale assesses levels of concern for falling while performing 16 different common tasks with the sum of scores ranging from 0-100, where 100 indicates [INSERT]. The Falls Efficacy Scale will be assessed pre- and post-intervention.
Change in Life-Space Assessment (LSA) Score | Baseline and 8 weeks
  The LSA is reported as the average weekly frequency and independence of life-space mobility, with a sum of scores ranging from 0-120, where higher scores indicate greater mobility. LSA will be measured pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan K McMahon, PhD, Principal Investigator — University of Minnesota School of Nursing
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No